CLINICAL TRIAL: NCT05102838
Title: Prospective Cohort Study on Prognosis of Patients With Hepatitis B/C in Hainan Province Danzhou City
Brief Title: Prospective Cohort Study on Prognosis of Patients With Hepatitis B/C
Status: Not yet recruiting | Type: Observational
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Lin Bingliang, Professor, Sun Yat-sen University
Other Study IDs: Spark Srudy
Record Dates: First submitted 2021-10-20; First posted 2021-11-02 (Actual); Last update posted 2021-11-02 (Actual); Status verified 2021-10

CONDITIONS: Hepatitis B; Hepatitis C
MeSH Terms: conditions — Hepatitis B; Hepatitis C

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples will be retained at each timepoints.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Hepatitis B cohort: 1. Patients with HBsAg and/or HBV DNA positive;
  2. Patients without cirrhosis.
  Interventions: Other: Anti-virus treatment
- Hepatitis C cohort: 1. Patients with anti-HCV and/or HCV RNA positive;
  2. Patients without cirrhosis.
  Interventions: Other: Anti-virus treatment
- Cirrhosis cohort: 1. Patients diagnosised with cirrhosis;
  2. Patients with HBsAg, and/or HBV DNA, and/or anti-HCV and/or HCV RNA positive.
  Interventions: Other: Anti-virus treatment
- Liver cancer cohort: 1. Patients diagnosised with liver cancer;
  2. Patients with HBsAg, and/or HBV DNA, and/or anti-HCV and/or HCV RNA positive.
  Interventions: Other: Anti-virus treatment

INTERVENTIONS:
Other: Anti-virus treatment — Anti-virus treatment

SUMMARY:
Hepatitis B (HBV) and hepatitis C (HCV) are prevalent all over the world, which seriously threatens public health. In 2016, the World Health Organization(WHO) put forward the goal of eliminating the threat of viral hepatitis to public health by 2030. However, at present, the diagnosis rate and treatment rate of chronic HBV and HCV in China are still far from the goal put forward by WHO. Therefore, for China, the elimination of viral hepatitis is still a public health problem that needs a long time to face.

This study aims to screen and follow up HBV and HCV patients in Danzhou City, Hainan Province, so as to understand the epidemiological characteristics and long-term prognosis of HBV/HCV patients.

DETAILED DESCRIPTION:
Hepatitis B (HBV) and hepatitis C (HCV) are prevalent all over the world, which seriously threatens public health. According to the survey, there are about 93 million chronic HBV infected people and 10 million chronic HCV infected people in China, accounting for 36.19% and 14.08% of the global HBV and HCV infected people respectively. Chronic HBV and HCV infection is the main cause of liver cirrhosis and liver cancer, which places a great burden on the national economy.

In 2016, the World Health Organization(WHO) put forward the goal of eliminating the threat of viral hepatitis to public health by 2030, including 90% diagnosis rate, 80% treatment rate and 90% cure rate of viral hepatitis, in order to reduce 65% of viral hepatitis related deaths and reduce the disease burden. However, at present, the diagnosis rate of chronic HBV in China is 18.7%, the treatment rate is 10.8%, the diagnosis rate of chronic HCV is 30%, and the treatment rate is 9%, which are still far from the goal put forward by WHO. Therefore, for China, the elimination of viral hepatitis is still a public health problem that needs a long time to face.

This study aims to screen and follow up HBV and HCV patients in Danzhou City, Hainan Province, so as to understand the epidemiological characteristics and long-term prognosis of HBV/HCV patients.

ELIGIBILITY:
Inclusion Criteria:

* HBsAg/HBV DNA positive
* or anti-HCV/HCV RNA positive

Exclusion Criteria:

* patients who refused to participate in the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Hepatitis B or hepatitis C patients will be enrolled in this study.
Sampling Method: Probability Sample
Enrollment: 60000 (Estimated)
Dates: Start 2021-11-01 (Estimated); Primary Completion 2025-08-30 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Epidemiological characteristics of hepatitis B and C | up to 192 weeks
  Epidemiological characteristics of hepatitis B and C in Danzhou City, Hainan Province
Long-term outcome | up to 192 weeks
  Long-term outcome of HBV/HCV infected patients in Danzhou City, Hainan Province
Risk factors | up to 192 weeks
  Risk factors for long-term outcome of HBV/HCV infected patients in Danzhou City, Hainan Province

SECONDARY OUTCOMES:
Incidence of cirrhosis | up to 192 weeks
  Incidence of cirrhosis for HBV/HCV infected patients in Danzhou City, Hainan Province
Incidence of liver cancer | up to 192 weeks
  ncidence of liver cirrhosis for HBV/HCV infected patients in Danzhou City, Hainan Province
Hepatic decompensation | up to 192 weeks
  Hepatic decompensation rate for HBV/HCV infected patients in Danzhou City, Hainan Province
Survival rate for liver cancer | up to 192 weeks
  Survival rate for liver cancer patients in Danzhou City, Hainan Province
Survival rate for cirrhosis | up to 192 weeks
  Survival rate for cirrhosis patients in Danzhou City, Hainan Province
HBV interruption rate of perinatal transmission | up to 192 weeks
  HBV interruption rate of perinatal transmission in Danzhou City, Hainan Province
HBsAg loss | up to 192 weeks
  The HBsAg loss rate of HBV infected patients in Danzhou City, Hainan Province

CONTACTS AND LOCATIONS:
Overall Officials: Bingliang Lin, Dr., Principal Investigator — Sun Yat-sen University

REFERENCES:
- [Background] 1.Lu FM, Zhuang H. Management of hepatitis B in China[J]. Chin Med J ( Engl) , 2009, 122(1): 3-4． 2.Chen YS, Li L, Cui FQ et al. Seroepidemiological study of hepatitis C in China[J].Chinese Journal of Epidemiology, 2011, 32:888-891. 3.Wang FS, Fan JG, Zhang Z, et al. The global burden of liver disease: the major impact of China[J]. Hepatology, 2014, 60(6): 2099 -2108． 4.Huang YW, Yang SS, Fu SC, et al. Increased risk of cirrhosis and its decompensation in chronic hepatitis C patients with new-onset diabetes: a nationwide cohort study[J]. Patology, 2014,60:807-814. 5.69th World Health Assembly. Draft Global Health Sector Strategies. April 2016. Available at: http://apps.who.int/gb/ebwha/pdf_files/WHA69/A69_32-en.pdf?ua=1 (accessed February 2017) 6.Global Hepatitis Report, 2017. http://www.who.int/mediacentre/factsheets/fs164/zh. 7.CDA Foundation's Polaris Observatory; 2020 Available from https://cdafound.org/polaris/ (Accessed 2020-06-09).